CLINICAL TRIAL: NCT03030092
Title: Maximal Strength Training Following Hip Fracture Surgery: Impact on Muscle Mass, Balance, Walking Efficiency and Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Berg10069
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Today's standard care
- Intervention group (Experimental): Maximal Strength Training
  Interventions: Other: Maximal Strength Training

INTERVENTIONS:
Other: Maximal Strength Training — leg pres and abduction exercises
  Arms: Intervention group

SUMMARY:
One group will receive today's standard rehabilitation program following hip fracture surgery. The intervention group will have maximal strength training incorporated in their program. It consists of 3 training sessions per week for 8 weeks, where 4-5 repetitions over 4 sets for leg press and abduction resistance exercise at ~85% of maximal strength is carried out. Muscle strength, balance and bone density will be compared between the groups following the 8-week rehabilitation period. The feasibility of the intervention for the patient group will be evaluated based on compliance with training program and possible adverse events related to the operated hip.

ELIGIBILITY:
Inclusion Criteria:

* age over 65, hip fracture surgery

Exclusion Criteria:

* COPD, Heart failure, Dementia

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 8 weeks
  1RM leg press, and hip abduction
Balance | 8 weeks
  unipedal stance test
Bone Density | 8 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134
- [Derived] Berg OK, Stutzer JM, Hoff J, Wang E. Early Maximal Strength Training Improves Leg Strength and Postural Stability in Elderly Following Hip Fracture Surgery. Geriatr Orthop Surg Rehabil. 2021 Apr 30;12:21514593211015103. doi: 10.1177/21514593211015103. eCollection 2021. PMID 34017617